CLINICAL TRIAL: NCT00921739
Title: Phase I Dose Escalation Study of Accelerated Fractionation With Esophageal Sparing Using Intensity-Modulated Radiation Therapy for Locally-Advanced Thoracic Malignancies Including a Prospective Assessment of Esophageal Motion and Radiation-Induced Esophageal Injury
Brief Title: Esophageal Sparing Intensity-modulated Radiation Therapy (IMRT) for Locally-Advanced Thoracic Malignancies
Acronym: ESIMRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00017361
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Cancer; Thymoma; Thymus Neoplasms
Keywords: Non small cell lung cancer; Small cell lung cancer; Thymoma unresectable; Thymic carcinoma unresectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thymoma; Thymus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT concurrent with chemotherapy (Experimental): 6 fractions of esophageal sparing IMRT weekly for 5-6 weeks (dependent on dose cohort) concurrent with standard chemotherapy: Cisplatin 50 mg/m2 /d intravenously (IV) on days 1, 8, 29, and 36. Etoposide 50 mg/m2 /d IV on days 1 through 5 and 29 through 33.
  Interventions: Radiation: Esophageal sparing IMRT

INTERVENTIONS:
Radiation: Esophageal sparing IMRT — 6 fractions/week of 2Gy each for 29 fx (58 Gy), 31 fx (62 Gy), 33 fx (66 Gy), 35 fx (70 Gy), or 37 fx (74 Gy).

SUMMARY:
Hypothesis 1- Using IMRT, the radiation therapy (RT) dose can be safely escalated from 58 Gy to 74 Gy given as 6 fractions/week with concurrent chemotherapy.

Hypothesis 2- Esophageal motion can be used to customize planning organ at risk volumes.

Hypothesis 3- Biological predictors of acute esophagitis can be used to identify patients at high risk of developing esophageal toxicity from radiation therapy and chemotherapy.

DETAILED DESCRIPTION:
Prospective phase I study designed to determine the maximum tolerated dose of radiation therapy given in an accelerated fashion (2 Gy/fraction, 6 fractions/week) with concurrent chemotherapy. Intensity-modulated radiation therapy (IMRT) will be utilized to spare the esophagus. All patients on the dose escalation study will participate in additional assessments evaluating esophageal motion and esophageal toxicity from radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of one of the following thoracic malignancies:

  * Non-small cell lung cancer (stage III or X (recurrent) with disease confined to local/regional sites)
  * Small cell lung cancer (stage II-III)
  * Thymoma (unresectable)
  * Thymic carcinoma (unresectable)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Weight loss < 10% in preceding 3 months prior to diagnosis
* ANC > or = 1500 and platelet count > or = 100,000.
* Creatinine clearance greater than 50 ml/min
* 18 years of age or older.
* Negative pregnancy test in women of child-bearing potential

Exclusion Criteria:

* Prior thoracic irradiation
* Medical contraindications to thoracic irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of IMRT | within 30 days of completing RT

SECONDARY OUTCOMES:
The occurrence of RT-induced acute esophagitis | One year
To determine if biological predictors of esophagitis can identify patients who develop severe esophageal toxicity during radiation therapy | Two years
  Blood will be drawn at specific time intervals, plasma will be analysed for Glutathione Oxidation, Citrulline, Lipid peroxidation, DNA oxidation, and Tetrahydrobiopterin.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelsey, MD, Principal Investigator — Duke University Medical Center, Dept Radiation Oncology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Socinski MA, Rosenman JG, Halle J, Schell MJ, Lin Y, Russo S, Rivera MP, Clark J, Limentani S, Fraser R, Mitchell W, Detterbeck FC. Dose-escalating conformal thoracic radiation therapy with induction and concurrent carboplatin/paclitaxel in unresectable stage IIIA/B nonsmall cell lung carcinoma: a modified phase I/II trial. Cancer. 2001 Sep 1;92(5):1213-23. doi: 10.1002/1097-0142(20010901)92:53.0.co;2-0. PMID 11571735
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Schild SE, Stella PJ, Geyer SM, Bonner JA, Marks RS, McGinnis WL, Goetz SP, Kuross SA, Mailliard JA, Kugler JW, Schaefer PL, Jett JR. Phase III trial comparing chemotherapy plus once-daily or twice-daily radiotherapy in Stage III non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):370-8. doi: 10.1016/s0360-3016(02)02930-9. PMID 12243810
- [Derived] Lafata KJ, Corradetti MN, Gao J, Jacobs CD, Weng J, Chang Y, Wang C, Hatch A, Xanthopoulos E, Jones G, Kelsey CR, Yin FF. Radiogenomic Analysis of Locally Advanced Lung Cancer Based on CT Imaging and Intratreatment Changes in Cell-Free DNA. Radiol Imaging Cancer. 2021 Apr;3(4):e200157. doi: 10.1148/rycan.2021200157. PMID 34114913